CLINICAL TRIAL: NCT01818284
Title: Plerixafor for Stem Cell Mobilization in Normal Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Proteonomix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0579; NCI-2013-02209 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-03-21; First posted 2013-03-26 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Blood And Marrow Transplantation
Keywords: Blood And Marrow Transplantation; Normal allogeneic donors; Stem cell mobilization; peripheral blood progenitor cells; PBPC; Allogeneic hematopoietic stem cell transplantation; HSCT; Donating blood stem cells; C-CSF; Neupogen; Filgrastim; Plerixafor; Mobozil; Apheresis
MeSH Terms: interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; plerixafor; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Filgrastim + Plerixafor (Experimental): Each donor receives Filgrastim 5 µg/kg subcutaneously in the morning daily for 4 days. The dose of Filgrastim based on the donor's actual body weight. Donors will continue Filgrastim until completion of apheresis. Each donor receives Plerixafor 240 µg/kg subcutaneously in the evening on the fourth day of Filgrastim mobilization. The dose-volume of Plerixafor based on the donor's actual body weight. Apheresis procedure to start the morning of day 5, approximately 10 to 11 hours after the administration of Plerixafor. The apheresis procedure will start in the morning of day 5, approximately 10 to 11 hours after the administration of Plerixafor.
  The apheresis procedure may continue beyond day 1 until the target dose of 4x106 cluster of differentiation 34 (CD34+) cells/kg (recipient's weight) is obtained.
  Interventions: Drug: Filgrastim; Drug: Plerixafor; Procedure: Apheresis Procedure

INTERVENTIONS:
Drug: Filgrastim — 5 µg/kg in the morning daily for 4 days.
  Other Names: Neupogen; Granulocyte-colony stimulating factor; G-CSF; GCSF; CSF-3
Drug: Plerixafor — 240 µg/kg subcutaneously in the evening on the fourth day of Filgrastim mobilization.
  Other Names: Mobozil
Procedure: Apheresis Procedure — The apheresis procedure will start in the morning of day 5, approximately 10 to 11 hours after the administration of Plerixafor.
  The apheresis procedure may continue beyond day 1 until the target dose of 4x106 CD34+ cells/kg (recipient's weight) is obtained.

SUMMARY:
The goal of this clinical research study is to learn if treating stem cell donors with filgrastim (G-CSF) and plerixafor (Mozobil®) can cause them to produce a higher number of blood stem cells than filgrastim by itself. Researchers also want to learn if giving both of these drugs helps donors produce enough stem cells so that only 1 apheresis procedure needs to be performed.

Researchers will study if using both drugs lowers the risk of the stem cell transplant recipients developing severe forms graft-versus-host disease (GVHD). GVHD is a condition in which transplanted tissue (such as blood stem cells) attacks the tissue of the recipient's body.

The safety and effectiveness of this drug combination will also be studied.

Filgrastim and plerixafor are both designed to help move or "mobilize" the stem cells from the bone marrow to the blood.

DETAILED DESCRIPTION:
Stem Cell Transplant:

You will receive blood stem cells from a donor on this study. You will sign a separate informed consent for the transplant procedure.

Follow-Up Visits:

About 1, 3, and 6 months after the transplant, an extra sample of bone marrow (about 2 teaspoons) will be collected at the same time as the standard of care bone marrow aspiration/biopsy procedures. This bone marrow sample will be tested to find out how well the donated stem cells have been accepted by your body. However, you will not have a separate bone marrow aspiration/biopsy only to collect bone marrow for this testing.

When you return to the clinic at 6, 9, and 12 months for routine transplant follow-up visits, the study staff will try to get information on your health status from the clinic notes in your medical record. If this is not possible, you may receive a phone call from the study staff to check your health status. These calls will last about 10 minutes.

Length of Treatment:

You will be on study for about 1 year after the transplant (including follow-up contact by phone, if needed).

You may be taken off study early if you are not able to follow study directions or if you decide to leave the study.

This is an investigational study. Filgrastim is FDA approved for use in stem cell collection. Plerixafor is FDA approved for use in patients with multiple myeloma and non-Hodgkin's lymphoma.

Up to 30 donor and recipient pairs will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Donor eligibility: Age >/= 10 years.
2. Donor eligibility: Related donors who met standard eligibility criteria and are willing to participate in this study.
3. Donor eligibility: Able to provide informed consent.
4. Recipient Eligibility: Patients who are scheduled to undergo an allogeneic related transplant and whose donors consented to participate in this study.
5. Recipient Eligibility: Able to provide informed consent.

Exclusion Criteria:

1) Donors who are on anti-coagulation or anti-platelet agents are not eligible.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chitra M. Hosing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 16, 2013 to May 1, 2015. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Filgrastim + Plerixafor for Donors: Filgrastim 5 µg/kg subcutaneously daily for 4 days until end of apheresis; Plerixafor 240 µg/kg subcutaneously on fourth day of Filgrastim mobilization; followed by Apheresis day 5 which may continue beyond day 1 until target dose of 4x10^6 CD34+ cells/kg (recipient's weight) obtained.
- Recipients: Recipients received Plerixafor mobilized cells for allogeneic hematopoietic stem cell transplantation (HSCT) on day 0 of their designated treatment plan (following day 5 of donor's Plerixafor study specific treatment plan).
Period: Overall Study
Arm/Group | Filgrastim + Plerixafor for Donors | Recipients
Started | 11 | 11
Completed | 7 | 5
Not Completed | 4 | 6
Not completed — Not eligible due to White Blood Counts | 4 | 4
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Donors Filgrastim + Plerixafor: Filgrastim 5 µg/kg subcutaneously daily for 4 days until end of apheresis; Plerixafor 240 µg/kg subcutaneously on fourth day of Filgrastim mobilization; followed by Apheresis day 5 which may continue beyond day 1 until target dose of 4x10^6 CD34+ cells/kg (recipient's weight) obtained.
- Recipients: Recipients received Plerixafor mobilized cells on day 0 of their designated treatment plan (following day 5 of donor's Plerixafor study specific treatment plan).
- Total: Total of all reporting groups
Arm/Group | Donors Filgrastim + Plerixafor | Recipients | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Median (Full Range); unit: years] | 58 [37 to 74] | 58 [41 to 71] | 58 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Summary of Most Common Toxicity: Donor Safety in Mobilizing Peripheral Blood Progenitor Cells (PBPC)
Description: Primary safety endpoint is the development of any unexpected toxicity (any grade 2 or higher non-hematologic toxicity) in donors. The severity of the toxicity - adverse events (AEs) graded according to Common Terminology Criteria v4.0 (CTCAE).
Time Frame: 5 days
Measure: Number; unit: adverse events
Groups:
- Donors: Filgrastim + Plerixafor: Filgrastim 5 µg/kg subcutaneously daily for 4 days until end of apheresis; Plerixafor 240 µg/kg subcutaneously on fourth day of Filgrastim mobilization; followed by Apheresis day 5 which may continue beyond day 1 until target dose obtained.
Arm/Group | Donors: Filgrastim + Plerixafor
Number analyzed (Participants) | 11
adverse events
  Tachycardia | 1
  Nausea | 2
  Insomnia | 2
  Bone pain | 2
  Injection site reaction | 1
  Diarrhea | 1
  Chest Pain | 1

2. Primary Outcome: Feasibility in Mobilizing PBPC in Donors: Number of Donors Reaching Stem Cell Target Collection on First Day of Collection Following Treatment of Filgrastim Plus Plerixafor
Description: Study determined to be feasible if all donors were able to receive Plerixafor without developing any grade 2 or higher non-hematologic toxicity. Feasibility of the combination of Filgrastim, Granulocyte-colony stimulating factor (G-CSF) plus Plerixafor is to effectively mobilize CD34+ cells so that an adequate transplant (>4 x 10^6 CD34+ cells/kg) can be reliably collected with one apheresis for allogeneic HSCT.
Time Frame: 4 days
Population: Four participants did not receive Plerixafor due to a white blood cell count outside of the protocol specific window. It should be noted, the protocol threshold for white blood cell count was amended from 40,000 to 45,000.
Measure: Count of Participants; unit: Participants
Arm/Group | Donors: Filgrastim + Plerixafor
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse event data collected for donors over one month period after first injection of filgrastim and for recipients from start of preparative regimen followed by infusion of allogeneic stem cell transplantation Day 0 to Day +30, up to 40 days.
Description: For the purpose of this study the treatment plan (preparative regimen followed by infusion of allogeneic stem cell transplantation) is defined as "transplant package"; therefore adverse events known to be caused by components of the transplant package and its direct consequences were collected.
Groups:
- Donors Filgrastim + Plerixafor: Filgrastim 5 µg/kg subcutaneously daily for 4 days until end of apheresis; Plerixafor 240 µg/kg subcutaneously on fourth day of Filgrastim mobilization; followed by Apheresis day 5 which may continue beyond day 1 until target dose of 4x106 CD34+ cells/kg (recipient's weight) obtained.
Arm/Group | Donors Filgrastim + Plerixafor | Recipients
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 5/11 | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donors Filgrastim + Plerixafor (N=11) | Recipients (N=11)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Mild tachicardia (Cardiac disorders) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 3 (3)
Nightsweats (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Elevated bilirubin (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neutropenic fever (Immune system disorders) | 0 (0) | 2 (2)
CMV Reactivation, Alpha-hemalytic streptococcus bacteremia (Infections and infestations) | 0 (0) | 2 (2)
Injection site reaction (Surgical and medical procedures) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (7)
Altered mental status related to pain medication (Nervous system disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Fluid Overload (Renal and urinary disorders) | 0 (0) | 1 (1)
Hand & foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Catheter related deep vein thrombosis (DTV) (Vascular disorders) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes